CLINICAL TRIAL: NCT05968508
Title: A Randomized, Double-blind, Single-dose, Two-arm Parallel Study to Compare the Pharmacokinetics and Safety of BAT1806 Prefilled Subcutaneous Injection With RoActemra® in Healthy Chinese Male Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bio-Thera Solutions (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: BAT-1806-003-CR
Record Dates: First submitted 2023-07-20; First posted 2023-08-01 (Actual); Last update posted 2025-05-29 (Actual); Status verified 2025-05

CONDITIONS: Healthy Men
MeSH Terms: interventions — tocilizumab

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- BAT1806 prefilled subcutaneous injection (Experimental)
  Interventions: Drug: BAT1806 prefilled subcutaneous injection/RoActemra® (from EU)
- RoActemra® (from EU) (Active Comparator)
  Interventions: Drug: BAT1806 prefilled subcutaneous injection/RoActemra® (from EU)

INTERVENTIONS:
Drug: BAT1806 prefilled subcutaneous injection/RoActemra® (from EU) — A total of 150 subjects are planned to be enrolled and 1:1randomized to receive single dose of 162 mg/0.9 mL BAT1806 injection, or RoActemra® (from EU) subcutaneously.

SUMMARY:
This is a randomized, double-blind, single-dose, two-arm parallel study to compare the pharmacokinetics, safety and immunogenicity of BAT1806 prefilled subcutaneous injection with RoActemra® (from EU) in healthy male subjects.

DETAILED DESCRIPTION:
A total of 150 subjects are planned to be enrolled and 1:1randomized to receive single dose of 162 mg/0.9 mL BAT1806 injection, or RoActemra® (from EU) subcutaneously.

A 14-day screening period is set in this study. Subjects will be admitted one day prior to administration (Day -1) and can be discharged only upon completion of relevant observations and evaluations after administration on Day 5. After discharge, subjects need to return to the hospital for 10 follow-ups as required in the study.

ELIGIBILITY:
Inclusion Criteria:

* Subjects can be enrolled only when they meet all the following inclusion criteria:

  1. Signed the informed consent form prior to the study, sufficient understanding of the content, procedure and possible adverse reactions of the study;
  2. Willing and able to comply with the visit and treatment specified in the study;
  3. Subjects (including their partners) who are willing to refrain from pregnancy, sperm donation and take effective contraceptive method in the future 6 months (i.e., 6 months after study medication), see Appendix 4 for the detailed contraceptive measures;
  4. Healthy male subjects aged 18～55 years (inclusive);
  5. BMI ranging from 18.0～28.0 kg/m2 (inclusive), and weight ranging from 55.0～85.0 kg (inclusive);
  6. Normal or abnormal physical examination that is judged as clinically insignificant;

Exclusion Criteria:

* Subjects can not be enrolled in this study if any of the following criteria is met:

  1. Smoking >5 cigarettes per day within three months prior to the study;
  2. Any serious allergic reaction to food or drug at present or in the past, or allergy to Tocilizumab, or serious allergy or allergic reaction to human, humanized or murine monoclonal antibody;
  3. History of excessive drinking (14 units of alcohol per week: 1 unit = 285 mL beer, or 25 mL liquor, or 125 mL wine);
  4. Blood donation or massive blood loss (>450 mL) within three months prior to screening, or plan for blood donation or surgery during the study;
  5. Intake of any prescription drug, over-the-counter drug, any vitamin product or herbal medicine within 28 days prior to screening;
  6. Great change in dietary or exercise habit within 2 weeks prior to screening or from screening to administration;
  7. Having any disease that may increase hemorrhagic risk, such as haemorrhoids with hemorrhagic symptoms, acute gastritis or gastric and duodenal ulcer;
  8. Clinically significant abnormality in echocardiography;
  9. Clinically significant abnormality in clinical laboratory examination, or other clinical findings showing the following disorders of clinical relevance (including but not limited to gastrointestinal, renal, hepatic, neurological, hematological, endocrine, oncological, pulmonary, immune, mental or cerebro- and cardiovascular diseases);
  10. Clinically significant (judged by investigators) abnormality in ECG, or QTcF > 450ms (allowed to be repeated for once, the subject needs to be excluded if the two measurements of QTcF are > 450ms);
  11. Acute disease or concomitant medication from screening to prior to administration of study drug;
  12. Positive urine drug screen, or history of drug abuse or use of narcotics in the past 5 years;
  13. Positive HBsAg in five hepatitis B markers at screening; or positive anti-HBc and negative anti-HBs; or positive hepatitis C antibody; or positive HIV antibody; or positive Treponema pallidum antibody;
  14. Intake of any alcohol-containing product within 48 hours prior to dosing of study drug, or failure to limit alcohol consumption as required during the study;
  15. Currently or previously having malignant tumor;
  16. History of hypertension, or systolic blood pressure ≥ 140 mmHg, or diastolic blood pressure ≥90 mmHg at screening/baseline (allowed to be repeated for once, the subject needs to be excluded if the two measurements of systolic blood pressure ≥ 140 mmHg, or diastolic blood pressure ≥90 mmHg);
  17. Patients with hepatic disorder who are judged by investigators as inappropriate for enrollment;
  18. Presence of active infection, including acute and chronic infection as well as local infection;
  19. Chest X-ray showing active pulmonary tuberculosis; or previous history of tuberculosis or latent tuberculosis infection, or clinical manifestations suspected as tuberculosis (including but not limited to pulmonary tuberculosis); Positive for T-SPOT®.TB interferon-γ-release assays, or contact with patients with tuberculosis within three months or/and symptoms or/and signs suspected as tuberculosis;
  20. Had received or plan to receive live virus vaccine or immunosuppressant within 12 weeks prior to administration of study drug;
  21. Having participated in drug clinical trial within three months prior to the first dose of study drug, or plan to participate in other drug clinical trial during the study;
  22. Those who are considered by investigators as inappropriate for enrollment.

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 300 (Actual)
Dates: Start 2023-08-29 (Actual); Primary Completion 2024-10-08 (Actual); Study Completion 2024-10-08 (Actual)

PRIMARY OUTCOMES:
AUC0-inf | from Day0 to Day57
AUC0-t | from Day0 to Day57
Cmax | from Day0 to Day57

CONTACTS AND LOCATIONS:
Overall Officials: Wei Hu, Ph.D, Principal Investigator — The Second Hospital of Anhui Medical University
Locations (1):
- The Second Affiliated Hospital of Anhui Medical University, Hefei, Anhui, China

REFERENCES:
- [Derived] Yang Q, Jiang Y, Liu Z, Wu J, Dong Q, Liu Y, Qin H, Zhang Q, Zhang Q, Hu W. A randomized, double-blind, single-dose, parallel two-group study comparing the pharmacokinetics, safety, and immunogenicity of BAT1806 SC with tocilizumab in healthy Chinese male subjects. Expert Opin Biol Ther. 2025 Oct;25(10):1101-1111. doi: 10.1080/14712598.2025.2574006. Epub 2025 Oct 14. PMID 41069221